CLINICAL TRIAL: NCT01849471
Title: Evaluation of Socioeconomic Aspects Before and After Primary Radiation Therapy (Percutaneous or Interstitial or Combined Percutaneous and Interstitial) in Patients With Prostate Cancer
Brief Title: Socioeconomic Aspects Before and After Radiation Therapy in Patient With Prostate Cancer
Acronym: ECOPRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: EP2013
Record Dates: First submitted 2013-04-18; First posted 2013-05-08 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: socioeconomic aspects; costs of therapy; follow-up costs; primary radiation; percutaneous; interstitial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with prostate cancer: questionnaires
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — patients receive questionnaires regarding socioeconomic aspects before, during and after therapy

SUMMARY:
This trial is an interrogation of patients with prostate cancer to evaluate socioeconomic effects of radiotherapy. Patients with percutaneous or interstitial or combined percutaneous and interstitial radiotherapy are included. Beside medical effects and adverse events, it's prospectively needed to extensively inform patients about socioeconomic aspects associated with radiotherapy. The interrogation comprises to collect possible costs and expenditures during and after therapy. Aspects especially concerning post therapy period include additional consultations, individual applied alternative medical care, need for additional medical aids (salves, medicine, bandages) and changes in professional and social situation. It's figured out in what extend costs are absorbed by health insurance coverage. In Germany there is no appropriate trial with respective patient population and respective therapy. Primary endpoint is the evaluation of therapy concerning and follow-up costs as well as changes in social and professional situation. Secondary endpoints are quality of life, adverse events of therapy and the correlation of quality of life, adverse events and economic aspects for the patient and the health insurance coverage.

ELIGIBILITY:
Inclusion Criteria:

* minimal age 18
* low, mediate and high-grade prostate cancer

Exclusion Criteria:

* tumor recurrence
* surgery as primary therapy
* prior radiotherapy except conventional radiotherapy
* patients with other malignancies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostata cancer that receive primary radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
therapy concerning and follow-up costs associated with changes in social professional situation that is connected with Quality of life | Participants will be followed for the duration of therapy and for 1 year after the last study treatment
  by questionnaires concerning social aspects and quality of life to evaluate connections between these parameters

SECONDARY OUTCOMES:
adverse events | Participants will be followed for the duration of therapy and for 1 year after the last study treatment
correlation of quality of life, adverse events and economic aspects for the patient and the health insurance coverage | Participants will be followed for the duration of therapy and for 1 year after the last study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annedore Strnad, MD, MHBA, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen; Rainer Fietkau, MD, Study Director — Strahlenklinik, Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Germany